CLINICAL TRIAL: NCT02502825
Title: Comparison of 2-min Tidal Breathing Methacholine Bronchial Provocation With Wright and Devilbiss646 Nebulizers
Brief Title: Comparison of Methacholine Bronchial Provocation With Wright and Devilbiss646 Nebulizers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Firestone Institute for Respiratory Health (Other)
Responsible Party: Principal Investigator, Jinping Zheng, deputy director, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GIRD201533
Record Dates: First submitted 2015-07-08; First posted 2015-07-20 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asthma (Experimental): methacholine(0.031-16mg/ml) bronchial provocation tests. this is a crossover,normal-control study. nebulized with Wright nebulizer for 2 minutes with an output of 0.13ml/min.
  Interventions: Other: methacholine; Device: Wright Nebulizer; Device: Devilbiss646 Nebulizer
- normal controls (Experimental): methacholine(0.031-16mg/ml) bronchial provocation tests. this is a crossover,normal-control study. nebulized with Devilbiss646 nebulizer for 2 minutes with an output of 0.13ml/min
  Interventions: Other: methacholine; Device: Wright Nebulizer; Device: Devilbiss646 Nebulizer

INTERVENTIONS:
Other: methacholine — methacholine (0.03,0.06,0.125,0.5,1.0,2.0,4.0,8.0,16.0 mg/ml),Canada
Device: Wright Nebulizer — nebulized for 2 minutes with an output of 0.13ml/min
Device: Devilbiss646 Nebulizer — nebulized for 2 minutes with an output of 0.13ml/min

SUMMARY:
The purpose of this study is to compare the diagnostic validity (sensitivity and specificity) and evaluate the safety of 2-min Tidal Breathing methacholine bronchial provocation tests with the Wright and Devilbiss646 nebulizers in asthmatic in Guangzhou.

DETAILED DESCRIPTION:
After screening,each asthmatic patient will visit the investigators' center 4 times.

During the first week, the patient will be randomised to undergo methacholine bronchial challenge with Wright or Devilbiss 646 nebulizer on two separate days, which are at least 24 hours but not more than 7 days apart.The above procedure will be repeated for each patient in one month. But the nebulizer will be selected in a reverse order.Provocative concentration induced a 20% decrease in forced expiratory volume in one second (PC20) will be calculated for each test. Record all the adverse events during the tests.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of asthma;
* stable for more than 4 weeks with FEV1≥65%pred

Exclusion Criteria:

* exacerbation within 3 months;
* upper airway infections within 4 weeks;
* concomitant of hypertension or heart diseases;
* pregnancy;
* under immunotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
percentage of the participants that tested positive to methacholine bronchial provocation with Wright or Devilbiss646 nebulizer | 5 minutes after each challenge

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events during the methacholine bronchial provocation tests with Wright nebulizer and Devilbiss646 nebulizer | during and until 5 minutes after each challenge

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, Principal Investigator — State Key Laboratory of Respiratory Disease; China Clinical Research Center of Respiratory Disease; First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China